CLINICAL TRIAL: NCT04276402
Title: Effect of Photobiomodulation by 808nm Diode Laser on the Stability of Orthodontic Mini-implants: A Randomized Clinical Split-Mouth Trial.
Brief Title: Effect of Photobiomodulation by 808nm Diode Laser on the Stability of Orthodontic Mini-implants.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Jacek Matys, Principal Investigator, Wroclaw Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WroclawMU3
Record Dates: First submitted 2020-02-14; First posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Malocclusion, Angle Class II
MeSH Terms: conditions — Malocclusion, Angle Class II | interventions — Lasers

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Right side of the maxilla (Experimental)
  Interventions: Procedure: Irradiation of implants with 808nm laser
- Left side of the maxilla (No Intervention)

INTERVENTIONS:
Procedure: Irradiation of implants with 808nm laser — Irradiation of implants with 808nm laser
  Arms: Right side of the maxilla

SUMMARY:
The study aimed to evaluate the influence of a 635nm diode laser on the stability of orthodontic mini-implants in vitro, as well as mini-implants failure rate (mini-implant loss) and patients pain level after the treatment. A randomized clinical split-mouth trial was concluded with 22 subjects (14 women, 8 men), 44 orthodontic mini-implants with a diameter 1.4mm and length of 10mm. Mini-implants were placed between teeth 3 and 4; and 13 and 14 (Universal Numbering System), in the area of the attached gingiva, 2 mm below mucogingival junction.

ELIGIBILITY:
Inclusion Criteria:

* patients with class II malocclusion defect requiring lateral maxillary teeth distillation based on the use of orthodontic mini-implant;
* the patients were treated first time using fixed orthodontic appliance;
* no systemic diseases;
* were not using anti-inflammatory drugs;

Exclusion Criteria:

* had used antibiotics in the previous 24 months;
* smokers;
* had history of radiotherapy,
* taking bisphosphonate medication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2019-07-05 (Actual); Primary Completion 2019-10-12 (Actual); Study Completion 2019-11-02 (Actual)

PRIMARY OUTCOMES:
stability of orthodontic mini-implants | 60 days
  The mini-implants stability was estimated employing a Periotest device (Medzintechnik Gulden e K, Modautal, Germany). The Periotest measurement system includes the sound formed from contact between an object and a metallic tapping bar in a handpiece, which is electromagnetically driven and electronically verified. The Periotest response detection is analyzed through a fast Fourier transform (FFT) algorithm. Simply put, the Periotest answer to tapping is estimated by an accelerometer and then analyzed. The signal generated by tapping is then transformed to a value called the Periotest value (PTV), which depends on the damping characteristics of the peri-implant tissue. The Periotest Test values (PTVs) are based on a numerical scale ranging from -8 to +50, defined by mathematical computation. The lower Periotest values indicate higher implant stability and thereupon the higher absorption effect of the target objects.

SECONDARY OUTCOMES:
Pain level (NRS scale) | 24 hours
  Each patient received a questionnaire for individual pain assessment (the numeric rating scale, NRS-11, grade level 0-10) immediately following placement of mini-implants. The maximum pain level was measured at both sides of the maxilla during the first day after the treatment. The NRS-11 scale consists of a conscious, subjective assessment of the pain experienced; therefore, it is used in the case of patients over ten years old.
  0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-10 = severe pain.
mini-implants loss | 60 days
  Mini-implants survival rate was assessed during 60 days observation period.

CONTACTS AND LOCATIONS:
Locations (1):
- Private Dental Healtcare, Kościan, Poland

IPD SHARING:
Plan to Share IPD: No